CLINICAL TRIAL: NCT03636464
Title: Pharmacokinetics and Deposition of Commonly Prescribed Antibiotics in Hospitalized Critically Ill Patients Undergoing Renal Replacement Therapies
Brief Title: Pharmacokinetics of Antibiotics in Patients Undergoing Renal Replacement Therapies
Acronym: RRTdose
Status: Recruiting | Type: Observational
Sponsor: Cleveland Clinic Abu Dhabi (Other)
Collaborators: University of the Sciences in Philadelphia (Other)
Responsible Party: Principal Investigator, Wasim El Nekidy, Senior Pharmacotherapy Specialist, Cleveland Clinic Abu Dhabi
Other Study IDs: A-2017-010
Record Dates: First submitted 2018-07-29; First posted 2018-08-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Renal Replacement Therapy
Keywords: Pharmacokinetics; antibiotics; RRT
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood collection — Pharmacokinetics

SUMMARY:
The study is aiming to describe the pharmacokinetic and pharmacodynamic profile of intravenous meropenem, ertapenem, cefepime, colistin, Ceftazidime/Avibactam , Ceftolozane/Tazobactam , and piperacillin/tazobactam in the plasma and determine how much is removed by Renal Replacement Therapies to ensure adequate dosing

DETAILED DESCRIPTION:
This pharmacokinetic evaluation and clinical outcomes will be an open-label study of 12-16 adult patients/antibiotic dose/modality to a total number of 180-240 patients, admitted to the acute care levels or intensive care unit at Cleveland Clinic Abu Dhabi receiving RRT and prescribed these seven antibiotics as recommended by their treating physicians. The collection of blood, ultrafiltrate or effluent fluids depending on RRT modality (HD or CRRT), and urine samples will begin after participants are administered first dose to determine if a loading dose will be required then after at least three doses (as prescribed by the treating physician) once these drugs will be at steady-state concentration. The study intervention duration will depend on dialysis modality expected to be 3 to 5 days depending on RRT modality and patients will be followed for outcomes (death or cure). Collected blood, effluent and urine samples will be assayed for drug concentration. The concentration data will be modeled by a computer program to determine the pharmacokinetic parameters used to predict future dosing in the case of RRT. Linear/logistic regression will be used as a component of statistical analysis to model the relationship between CRRT machine settings and the amount of the study drugs that will be removed by the filter. Information related to adverse events , clinical and microbiological cure will be collected in case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 year old
* Prescribed meropenem, ertapenem, cefepime, colistin, Ceftazidime/Avibactam , Ceftolozane/Tazobactam , or piperacillin/tazobactam for treatment of infection as part of standard medical care
* Administered meropenem, ertapenem, cefepime, colistin, Ceftazidime/Avibactam , Ceftolozane/Tazobactam ,or piperacillin/tazobactam while on renal replacement therapy (IHD or CRRT) or renal replacement therapy started while on any of these antibiotics
* Patients with hemoglobin > 70 g/L without blood transfusion in the past 24 hours
* Informed consent given by patient, next of kin or legally authorized representative

Exclusion Criteria:

* Less than 18 years of age
* Pregnant females
* Body mass index < 18 or > 35 kg/m2
* Presence of anemia (defined as hemoglobin < 70 g/L), thrombocytopenia, or leukopenia as defined by hematocrit, platelet, or white blood cell count < 75% of the lower limit of normal
* Concomitant receipt of another cephalosporin interfering with assay
* Participants likely to require surgical interventions during the study period if the surgery would interfere with dosing intervals or affect sampling process
* Protected patients; prisoners, patients with HIV, patients with physical or mental disabilities, psychiatric patients.
* Patients with documented life-threatening allergy (i.e anaphylaxis, angioedema) to any of the study drugs or their class.
* Patients with conditions known to significantly affect PK; (i.e. severe burn, significant ascites, spinal cord injury and cystic fibrosis)
* Any other reason felt by the investigators to potentially affect the outcomes of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on renal replacement therapy, prescribed antibiotics in the regular course of care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Serum antibiotic concentrations over time during dose interval | 24 months
  Blood will be collected at designated time points, serum samples will be assayed for drug concentration over time to describe pharmacokinetic disposition

SECONDARY OUTCOMES:
Amount of antibiotic removed by dialysis | 24 months
  Dialysate will be collected and assayed for drug concentration to determine the amount of drug cleared by RRT with respect to different dialysis modalities and membranes
Time above minimum inhibitory concentration (T/MIC) for time dependent antibiotics | 24 months
  Concentration/time data will be modeled mathematically (population pharmacokinetics and Monte Carlo simulation) to identify adequate dosing in this patient population
Area under concentration time curve over minimum inhibitory concentration for (Cmax/MIC) for concentration dependent antibiotics | 24 months
  Concentration/time data will be modeled mathematically (population pharmacokinetics and Monte Carlo simulation) to identify adequate dosing in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Wasim El Nekidy, PharmD, Principal Investigator — Cleveland Clinic Abu Dhabi; Islam Ghazi, PharmD, Principal Investigator — University of the Sciences
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided